CLINICAL TRIAL: NCT02143765
Title: An Open, Multi-center, Randomized Study to Evaluate the Efficacy and Safety of Mitiglinide Versus Acarbose in Patients With Type 2 Diabetes Mellitus in China
Brief Title: Efficacy and Safety of Mitiglinide vs Acarbose in Patients With Type 2 Diabetes Mellitus
Acronym: Match-101
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Zilin Sun, Chief of Department of Endocrinology, Zhongda Hospital, Institute of Diabetes, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhongdaH-Match
Record Dates: First submitted 2014-05-03; First posted 2014-05-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Mitiglinide; Acarbose; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitiglinide; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitiglinide (Experimental): Mitiglinide 10 mg three times a day, orally, for 12 weeks
  Interventions: Drug: Mitiglinide
- Acarbose (Active Comparator): Acarbose 50 mg three times a day, orally, for 12 weeks
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Mitiglinide — three times a day, orally, for 12 weeks
  Other Names: FADI
  Arms: Mitiglinide
Drug: Acarbose — three times a day, orally, for 12 weeks
  Other Names: PRECOSE
  Arms: Acarbose

SUMMARY:
Mitiglinide, a benzylsuccinic acid derivative, exerts selective action on the ATP-dependent K (KATP) channel of pancreatic β-cells and reportedly possesses a stronger affinity to the channel compared with other insulinotropic sulphonylurea receptor ligands, namely repaglinide and nateglinide. Preprandial administration of mitiglinide efficiently reduces postprandial hyperglycemia and improves overall glycemic control.

This was a 12-week, open, randomized study for comparing Mitiglinide versus Acarbose. The purpose of this study is to evaluate the efficacy and safety of Mitiglinide vs Acarbose in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Group I (Mitiglinide): Mitiglinide 10 mg three times a day, orally, for 12 weeks Group II (Acarbose): Acarbose 50 mg three times a day, orally, for 12 weeks Total subjects: 248, randomized to 2 groups at ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 70, regardless of gender
2. Subjects with type-2 diabetes mellitus diagnosed according to 1999 WHO criteria within 5 years
3. Subjects who had not received insulin secretagogues, insulin sensitizers, incretin mimetics or alpha-glucosidase inhibitors
4. Subjects whose fasting blood glucose [FBG] between7.0 and10.0 mmol/L and HbA1c ratio is between 7.0% and 10.0%

Note: Incretin mimetics contain glucagon-like peptide 1 (GLP-1) receptor agonist (including GLP-1 analogues) and dipeptidyl peptidase 4 inhibitors.

Exclusion Criteria:

1. Subjects with abnormal hepatic function whose aspartate transaminase (AST) and alanine transaminase (ALT) are 2 times higher than the upper limits of normal (ULN)
2. Subjects with renal disfunction whose plasma creatinine concentration are more than 1.1 ULN or positive urine protein
3. Subjects with severe heart disease, liver diseases, kidney disease and other serious organic disease
4. Subjects who have chronic intestinal diseases associated with marked disorders of digestion or absorption and may deteriorate as a result of increased gas formation in the intestine (like Gastrocardiac Syndrome, severe hernia, intestinal obstruction, intestinal ulcer and intestinal surgery)
5. Subjects with endocrine system diseases such as hyperthyroidism and cushing's syndrome etc.
6. Subject is contraindicated or hypersensitivity to both experimental drugs or comparator drugs
7. Subjects who participated in other clinical studies as subjects within 3 months before this study
8. Female subjects who have been pregnant , lactating or without contraception in childbearing potential
9. Subjects judged unfit for this study by investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12 | Baseline and Week 12

SECONDARY OUTCOMES:
the change from baseline to the end of treatment in fasting blood glucose (FBG), postprandial blood glucose (PBG) | Baseline, 4 weeks, 8 weeks, 12 weeks
Number of Participants with Serious and Non-Serious Adverse Events | up to 12 weeks
  Adverse events will be collected and followed in order to evaluate safety and tolerability
the change from baseline to the end of treatment in Diabetes Quality of Life | baseline and 12 weeks
  measured by Diabetes specific Quality of Life scale (DSQL) at baseline and 12 weeks
Treatment compliance | up to 12 weeks
Diabetes Treatment Satisfaction | 12 weeks
  measured by Diabetes Treatment Satisfaction Questionnaire (DTSQs) at 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second People's Hospital of Huai'an, Huai'an, Jiangsu
  - Department of Endocrinology, Zhongda Hospital, Institute of Diabetes, Southeast University, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Yancheng City No.1 People's Hospital, Yancheng, Jiangsu
  - Zhenjiang First People's Hospital, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] LV Xiaofeng. Clinical study on efficacy and safety of mitiglinide on type 2 diabetes mellitus. Chinese Journal of Clinical Pharmacology and Therapeutics, 2009, 14(2):175-179.
- [Result] Zhu Q, Tong Y, Wu T, Li J, Tong N. Comparison of the hypoglycemic effect of acarbose monotherapy in patients with type 2 diabetes mellitus consuming an Eastern or Western diet: a systematic meta-analysis. Clin Ther. 2013 Jun;35(6):880-99. doi: 10.1016/j.clinthera.2013.03.020. Epub 2013 Apr 18. PMID 23602502